CLINICAL TRIAL: NCT06337851
Title: Comparing Simultaneous and Consecutive Drainage of Bilateral Chronic Subdural Hematoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hasan Kamil Sucu, Neurosurgeon, Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AtaturkTRH2003/9
Record Dates: First submitted 2024-01-20; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Subdural Hematoma, Chronic
Keywords: Drainage; Chronic Subdural Hematoma; Consecutive; Simultaneous
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Intervention Model Description: a prospective randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous burr hole craniostomy (Group-1) (Active Comparator): Patients in group-1 were fixed in supine position with their heads in neutral and flexion position. Bilateral burr holes were made one after another, the dural surfaces were exposed at the same time, then the outer membranes of both sides opened and hematomas evacuated simultaneously. All the patients underwent a drainage system, performed with the insertion of a silicone tube into the subdural space and tunneled under the scalp to the exit point.
  Interventions: Other: Simultaneous burr hole craniostomy
- Consecutive burr hole craniostomy (Group-2) (Active Comparator): In group-2, hematoma with a greater thickness was removed first (if thickness was equal on both sides, first incision was made on the right side). The head in supine position was rotated to the side with a smaller hemorrhage thickness. Previously, burr holes were made, the dural surfaces were exposed, the outer membrane opened, and the hematoma was evacuated at one side. Then, drainage system inserted into the subdural space. After the procedure of the first side was completed, as a consecutive process, the head was rotated to the other side, and the same procedure was repeated.
  Interventions: Other: Consecutive burr hole craniostomy

INTERVENTIONS:
Other: Simultaneous burr hole craniostomy — Patients in group-1 were fixed in supine position with their heads in neutral and flexion position. Bilateral burr holes were made one after another, the dural surfaces were exposed at the same time, then the outer membranes of both sides opened and hematomas evacuated simultaneously. All the patients underwent a drainage system, performed with the insertion of a silicone tube into the subdural space and tunneled under the scalp to the exit point.
  Arms: Simultaneous burr hole craniostomy (Group-1)
Other: Consecutive burr hole craniostomy — In group-2, hematoma with a greater thickness was removed first (if thickness was equal on both sides, first incision was made on the right side). The head in supine position was rotated to the side with a smaller hemorrhage thickness. Previously, burr holes were made, the dural surfaces were exposed, the outer membrane opened, and the hematoma was evacuated at one side. Then, drainage system inserted into the subdural space. After the procedure of the first side was completed, as a consecutive process, the head was rotated to the other side, and the same procedure was repeated. The contralateral hematoma was evacuated.
  Arms: Consecutive burr hole craniostomy (Group-2)

SUMMARY:
Surgical evacuation CSDH via burr hole craniostomy appears to be the most widely practiced treatment technique worldwide and outcomes are generally favorable.

In previous reports, bilateral CSDH was raised as a predictor of rapid deterioration and worse outcomes attributable to brain herniation, in comparison with unilateral ones. Nevertheless, the optimal surgical considerations in bilateral CSDH still remain controversial. Thus, this study principally aims to finding out whether consecutive removal of bilateral CSDH really poses a complication risk. The secondary objectives of the study were to obtain information about the one-year prognosis of bilateral CSDH and to find factors that affect the prognosis, if any.

Inclusion criteria Symptomatic adult (≥18 years-old) patients with bilateral hemispheric CSDH

Exclusion criteria Patients with hematoma thickness smaller than 10 mm on either side, and those who previously underwent any cranial surgery

Randomization Simple randomization, without blocking, will be used to divide patients into two groups simultaneous burr hole craniostomy (Group-1) and consecutive burr hole craniostomy (Group-2).

Clinical Evaluation Neurological examination and scoring systems (Glasgow coma scale and Markwalder Grading) will be used.

Radiological Evaluation Radiological evaluations will be made with CT and MR imaging.

Operation Patients in group-1 were fixed in supine position with their heads in neutral and flexion position. Bilateral burr holes were made one after another, the dural surfaces were exposed at the same time, then the outer membranes of both sides opened and hematomas evacuated simultaneously. All the patients underwent a drainage system, performed with the insertion of a silicone tube into the subdural space and tunneled under the scalp to the exit point. In group-2, hematoma with a greater thickness was removed first (if thickness was equal on both sides, first incision was made on the right side). The head in supine position was rotated to the side with a smaller hemorrhage thickness. Previously, burr holes were made, the dural surfaces were exposed, the outer membrane opened, and the hematoma was evacuated at one side. Then, drainage system inserted into the subdural space. After the procedure of the first side was completed, as a consecutive process, the head was rotated to the other side, and the same procedure was repeated. The contralateral hematoma was evacuated.

Follow-Up Depending on the subdural fluid collected, all drains will be removed within post-operative 36-48 hours.

Only the patients with epileptic history and on epileptic medication will receive postoperative antiepileptics.

In the postoperative period, a comprehensive evaluation encompassing neurological examinations and CT imaging will be performed.

This evaluation protocol will be executed immediately following the surgical procedure, after the removal of surgical drains (usually on the second postoperative day), and at designated intervals of the 1st, 3rd, 6th, and 12th months to monitor patient progress and recovery.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) arises at the dural border cell layer and is characterized by a pathological collection of blood, fibrin, and degradation products between the dura mater and the arachnoid mater with an insidious onset and progression. Surgical evacuation CSDH via burr hole craniostomy appears to be the most widely practiced treatment technique worldwide and outcomes are generally favorable.Although unilateral CSDH is seen in the majority of patients, bilateral involvement is not rare in neurosurgical practices.

In previous reports, bilateral CSDH was raised as a predictor of rapid deterioration and worse outcomes attributable to brain herniation, in comparison with unilateral ones. Nevertheless, the optimal surgical considerations in bilateral CSDH still remain controversial. Thus, this study principally aims to finding out whether consecutive removal of bilateral CSDH really poses a complication risk. The secondary objectives of the study were to obtain information about the one-year prognosis of bilateral CSDH and to find factors that affect the prognosis, if any.

The study is conducted as a prospective randomized controlled trial.

Inclusion criteria Symptomatic adult (≥18 years-old) patients with bilateral hemispheric CSDH

Exclusion criteria Patients with hematoma thickness smaller than 10 mm on either side, and those who previously underwent any cranial surgery will be excluded.

Randomization Simple randomization, without blocking, will be used to divide patients into two groups simultaneous burr hole craniostomy (Group-1) and consecutive burr hole craniostomy (Group-2). Written consent will be taken from each patient and/or patient's relatives for the surgery and the use of data for this study.

Clinical Evaluation Neurological examination and scoring systems (Glasgow coma scale and Markwalder Grading) will be used.

Radiological Evaluation Radiological evaluations will be made with CT and MR imaging.

Operation The patients were operated on either under general or local anesthesia based on the recommendations of anesthesiologists and the patient's general medical status. First-generation cephalosporins were used as preoperative prophylactic antibiotics (cefazolin). Patients in group-1 were fixed in supine position with their heads in neutral and flexion position. Bilateral burr holes were made one after another, the dural surfaces were exposed at the same time, then the outer membranes of both sides opened and hematomas evacuated simultaneously. All the patients underwent a drainage system, performed with the insertion of a silicone tube into the subdural space and tunneled under the scalp to the exit point. In group-2, hematoma with a greater thickness was removed first (if thickness was equal on both sides, first incision was made on the right side). The head in supine position was rotated to the side with a smaller hemorrhage thickness. Previously, burr holes were made, the dural surfaces were exposed, the outer membrane opened, and the hematoma was evacuated at one side. Then, drainage system inserted into the subdural space. After the procedure of the first side was completed, as a consecutive process, the head was rotated to the other side, and the same procedure was repeated. The contralateral hematoma was evacuated. 12-gauge soft drainage sets with secretion bags were used for postoperative drainage in both groups.

Follow-Up Depending on the subdural fluid collected, all drains will be removed within post-operative 36-48 hours.

Only the patients with epileptic history and on epileptic medication will receive postoperative antiepileptics.

In the postoperative period, a comprehensive evaluation encompassing neurological examinations and CT imaging will be performed.

This evaluation protocol will be executed immediately following the surgical procedure, after the removal of surgical drains (usually on the second postoperative day), and at designated intervals of the 1st, 3rd, 6th, and 12th months to monitor patient progress and recovery.

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic bilateral hemispheric CSDH

Exclusion Criteria:

* Hematoma thickness smaller than 10 mm on either side
* Previously underwent any cranial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The Primary Outcome: Mortality | Postoperative first 12 months
  As the Primary Outcome, we considered the success of the operation at the end of the 12-month control period (we considered patients who died or were reoperated as unsuccessful).
The Primary Outcome: Early Postoperative Success Rate (Redo Surgery) | Postoperative first 12 months
  As the Primary Outcome, we considered the success of the operation at the end of the 12-month control period (we considered patients who died or were reoperated as unsuccessful).

SECONDARY OUTCOMES:
The secondary outcome: Follow-up assessment (Age) | One-year
  The impact of age on the one-year prognosis of bilateral chronic subdural hematoma was assessed.
The secondary outcome: Follow-up assessment (Sex) | One-year
  The impact of sex on the one-year prognosis of bilateral chronic subdural hematoma was assessed.
The secondary outcome: Follow-up assessment (Trauma-Relation) | One-year
  The impact of trauma-relation on the one-year prognosis of bilateral chronic subdural hematoma was assessed.
The secondary outcome: Follow-up assessment (Concomitant Pathologies) | One-year
  The impact of concomitant pathologies on the one-year prognosis of bilateral chronic subdural hematoma was assessed.
The secondary outcome: Follow-up assessment (The Glasgow Coma Scale) | One-year
  The assessment aimed to determine whether the Glasgow Coma Scale scores at each follow-up period had an impact on the prognosis of bilateral chronic subdural hematoma. The Glasgow Coma Scale is reported as the combined score (which ranges from 3 to 15) and the score of each test (E for eye from 1 to 4, V for Verbal from 1 to 5, and M for Motor from1 to 6). Higher score indicates better result.
The secondary outcome: Follow-up assessment (The Markwalder Grading Scale) | One-year
  The assessment aimed to determine whether the Markwalder Grading Scale scores at each follow-up period had an impact on the prognosis of bilateral chronic subdural hematoma.
  0: Patient neurological normal
  1. Patient alert and oriented; mild symptoms such as headache; absent or mild neurological deficit such as reflex asymmetry
  2. Patient drowsy (defined as Glasgow Coma Scale (GCS) score: 13-14) or disoriented with variable neurological deficit, such as hemiparesis
  3. Patient stuporous (defined as GCS 9-12) but responding appropriately to noxious stimuli; severe focal signs such as hemiplegia
  4. Patient comatose (GCS 8 or lower) with absent motor responses to painful stimuli; decerebrate or decorticate posturing.
The secondary outcome: Follow-up assessment (Neurological Examination - Motor) | One-year
  The assessment aimed to determine whether the neurological examination (motor lateraling findings) at each follow-up period had an impact on the prognosis of bilateral chronic subdural hematoma. --Motor deficit present or absent.
The secondary outcome: Follow-up assessment (Neurological Examination - fundus oculi) | One-year
  The assessment aimed to determine whether the neurological examination (fundus oculi examination) at each follow-up period had an impact on the prognosis of bilateral chronic subdural hematoma. -- papilledema present or absent.
The secondary outcome: Follow-up assessment (Neurological Examination - babinski sign) | One-year
  The assessment aimed to determine whether the neurological examination (Babinski's Sign) at each follow-up period had an impact on the prognosis of bilateral chronic subdural hematoma. Babinski sign present or absent.
The secondary outcome: Follow-up assessment (Radiological Assessments - midline shift) | One-year
  It was evaluated whether radiological assessment findings (midline shift) affected the prognosis of bilateral CSDH. -- length measurement in mm
The secondary outcome: Follow-up assessment (Radiological Assessments - hematoma volum) | One-year
  It was evaluated whether radiological assessment findings (hematoma volume) affected the prognosis of bilateral CSDH. -- volume measurement in cm3

CONTACTS AND LOCATIONS:
Overall Officials: Omer Akar, MD, Principal Investigator — Izmir Ataturk Training and Research Hospital
Locations (1):
- Izmir Ataturk Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the International Clinical Trials Registration Platform (ICTRP) became operational in 2007 and we do not have such a clinical trial registry system at the national level, the registration was made retrospectively. The first surgery date of the last patient included in the study was January 2004, and the recruitment period lasted approximately 6.5 years. This policy applies to trials that began enrolling participants on or after January 1, 2019.

REFERENCES:
- [Background] Okuchi K, Fujioka M, Maeda Y, Kagoshima T, Sakaki T. Bilateral chronic subdural hematomas resulting in unilateral oculomotor nerve paresis and brain stem symptoms after operation--case report. Neurol Med Chir (Tokyo). 1999 May;39(5):367-71. doi: 10.2176/nmc.39.367. PMID 10481440
- [Background] Kurokawa Y, Ishizaki E, Inaba K. Bilateral chronic subdural hematoma cases showing rapid and progressive aggravation. Surg Neurol. 2005 Nov;64(5):444-9; discussion 449. doi: 10.1016/j.surneu.2004.12.030. PMID 16253697
- [Background] Huang YH, Yang KY, Lee TC, Liao CC. Bilateral chronic subdural hematoma: what is the clinical significance? Int J Surg. 2013;11(7):544-8. doi: 10.1016/j.ijsu.2013.05.007. Epub 2013 May 24. PMID 23707986
- [Background] Agawa Y, Mineharu Y, Tani S, Adachi H, Imamura H, Sakai N. Bilateral Chronic Subdural Hematoma is Associated with Rapid Progression and Poor Clinical Outcome. Neurol Med Chir (Tokyo). 2016;56(4):198-203. doi: 10.2176/nmc.oa.2015-0256. Epub 2016 Feb 29. PMID 26923835
- [Background] Sucu HK, Gokmen M, Ergin A, Bezircioglu H, Gokmen A. Is there a way to avoid surgical complications of twist drill craniostomy for evacuation of a chronic subdural hematoma? Acta Neurochir (Wien). 2007 Jun;149(6):597-9. doi: 10.1007/s00701-007-1162-9. Epub 2007 May 7. PMID 17486289
- [Background] Nakaguchi H, Tanishima T, Yoshimasu N. Relationship between drainage catheter location and postoperative recurrence of chronic subdural hematoma after burr-hole irrigation and closed-system drainage. J Neurosurg. 2000 Nov;93(5):791-5. doi: 10.3171/jns.2000.93.5.0791. PMID 11059659
- [Background] Gokmen M, Sucu HK, Ergin A, Gokmen A, Bezircio Lu H. Randomized comparative study of burr-hole craniostomy versus twist drill craniostomy; surgical management of unilateral hemispheric chronic subdural hematomas. Zentralbl Neurochir. 2008 Aug;69(3):129-33. doi: 10.1055/s-2007-1004587. Epub 2008 Jul 29. PMID 18666056
- [Background] Markwalder TM, Steinsiepe KF, Rohner M, Reichenbach W, Markwalder H. The course of chronic subdural hematomas after burr-hole craniostomy and closed-system drainage. J Neurosurg. 1981 Sep;55(3):390-6. doi: 10.3171/jns.1981.55.3.0390. PMID 7264730
- [Background] Yagnik KJ, Goyal A, Van Gompel JJ. Twist drill craniostomy vs burr hole drainage of chronic subdural hematoma: a systematic review and meta-analysis. Acta Neurochir (Wien). 2021 Dec;163(12):3229-3241. doi: 10.1007/s00701-021-05019-3. Epub 2021 Oct 14. PMID 34647183
- [Background] Kolias AG, Chari A, Santarius T, Hutchinson PJ. Chronic subdural haematoma: modern management and emerging therapies. Nat Rev Neurol. 2014 Oct;10(10):570-8. doi: 10.1038/nrneurol.2014.163. Epub 2014 Sep 16. PMID 25224156